CLINICAL TRIAL: NCT00163215
Title: Evolution Of Growth Rate In Children Suffering From A Disease Associated With Growth Retardation and Treated By Genotonorm. A Pilot Study.
Brief Title: Growth Retardation In Children With Special Pathological Conditions Or Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6281269
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Results first posted 2012-12-19 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-11

CONDITIONS: Endocrine System Diseases
MeSH Terms: conditions — Endocrine System Diseases | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Somatropin (Experimental)
  Interventions: Drug: Somatropin

INTERVENTIONS:
Drug: Somatropin — Adapted dosage based on IGF 1 level and weight Form: liquid; Dosage and Frequency: from 0.0033mg/kg/day to 0.0067 mg/kg/day; Duration: 3 years

SUMMARY:
To show an increase in annual growth rate 3 years after Visit 2. Annual growth rate in standard deviation (SD) after 3 years will be compared to growth rate before the start of GH treatment.

ELIGIBILITY:
Inclusion Criteria:

* Bone age < 13 years for a boy and < 11 years for a girl
* Naive child: Measured Height < -2.5 SD for CA
* Child currently treated by GH

Exclusion Criteria:

* Idiopathic short stature
* Syndrome known to be associated with an increased risk of cancer e.g. family history of adenomatous polyposis

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2005-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- France (14):
  - Pfizer Investigational Site, Annemasse
  - Pfizer Investigational Site, Besançon
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Bron
  - Pfizer Investigational Site, Dijon
  - Pfizer Investigational Site, Grenoble
  - Pfizer Investigational Site, Lorient
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Pringy
  - Pfizer Investigational Site, Toulouse
  - Pfizer Investigational Site, Vandœuvre-lès-Nancy

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6281269&StudyName=Growth%20Retardation%20In%20Children%20With%20Special%20Pathological%20Conditions%20Or%20Disease%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Genotonorm: Genotonorm (recombinant somatropin) up to maximum of 50 microgram/kilogram/day (mcg/kg/day) subcutaneously as decided by the investigator, divided in 7 daily doses for up to 3 years.
Period: Overall Study
Arm/Group | Genotonorm
Started | 46
Completed | 31
Not Completed | 15
Not completed — Lack of Efficacy | 3
Not completed — Withdrawal by Subject | 5
Not completed — Other | 7

BASELINE CHARACTERISTICS:
Arm/Group | Genotonorm
Number analyzed (Participants) | 46
Age Continuous [Mean (Standard Deviation); unit: years] | 10.3 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 34

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Annual Growth Rate Standard Deviation Score (SDS) for Chronological Age (CA) at Month 36 in Intent-to-Treat (ITT) Population
Description: Change in annual growth rate (AGR) standard deviation score (SDS) for chronological age (CA) derived by subtracting AGR SDS CA at baseline from each time point (Yx) value. AGR at Yx= (height Yx-height Y[x-1])/([date of Yx-date of Y{x-1}]/365.25). AGR as SDS calculated using Sempe reference means and standard deviations (SD) for growth rate. AGR SDS CA (for both baseline and Yx)= (AGR-reference mean for growth rate CA)/reference SD for growth rate CA. CA calculated as integer (Date of height measurement-Date of birth)/365.25*12. SDS indicates how similar participant was to reference population.
Time Frame: Baseline, Month 36
Population: Intent to Treat (ITT) set included all participants who received at least 1 dose of study medication and had at least 1 evaluation of height after start of study medication. Here 'N' (Number of participants analyzed) signifies those participants who were evaluable for this measure and "n" signifies participants evaluated at that time point.
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Genotonorm
Number analyzed (Participants) | 42
SDS
  Baseline (n = 42) | -1.29 (1.79)
  Change at Month 36 (n = 26) | 2.36 (1.98)

2. Primary Outcome: Change From Baseline in Annual Growth Rate Standard Deviation Score (SDS) for Chronological Age (CA) at Month 36 in Per-Protocol (PP) Population
Description: as for outcome 1
Time Frame: Baseline, Month 36
Population: Per Protocol (PP) analysis set included all participants in the ITT set without a major protocol violation. Here 'N' (Number of participants analyzed) signifies those participants who were evaluable for this measure and "n" signifies participants evaluated at that time point.
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Genotonorm
Number analyzed (Participants) | 14
SDS
  Baseline (n = 14) | -1.98 (1.06)
  Change at Month 36 (n = 12) | 2.70 (2.02)

3. Secondary Outcome: Change From Baseline in Annual Growth Rate at Month 12, Month 24 and Month 36 in ITT Population
Description: Change in AGR at Yx was derived by subtracting AGR at baseline from Yx value. Annual growth rate was calculated each year and rescaled to 1 year if the interval between Yx and Y[x-1] was not 365 days, as long as a participant remained in the study. AGR at Yx was calculated using the previous height measurements (Y[x-1]) and height recorded at Yx (AGR Yx = [height Yx-height Y{x-1}] / ([date of Yx - date of Y{x-1}] /365.25).
Time Frame: Baseline, Month 12, Month 24, Month 36
Population: ITT set included all participants who received at least 1 dose of study medication and had at least 1 evaluation of height after start of study medication. Here 'N' (Number of participants analyzed) signifies those participants who were evaluable for this measure and "n" signifies participants evaluated at that time point.
Measure: Mean (Standard Deviation); unit: centimeter per year (cm/year)
Arm/Group | Genotonorm
Number analyzed (Participants) | 42
centimeter per year (cm/year)
  Baseline (n = 42) | 4.5 (1.8)
  Change at Month 12 (n = 36) | 3.3 (2.9)
  Change at Month 24 (n = 35) | 2.5 (2.7)
  Change at Month 36 (n = 26) | 2.0 (2.0)

4. Secondary Outcome: Change From Baseline in Annual Growth Rate at Month 12, Month 24, Month 36 in PP Population
Description: as for outcome 3
Time Frame: Baseline, Month 12, Month 24, Month 36
Population: PP analysis set included all participants in the ITT set without a major protocol violation. Here 'N' (Number of participants analyzed) signifies those participants who were evaluable for this measure and "n" signifies participants evaluated at that time point.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Genotonorm
Number analyzed (Participants) | 14
cm/year
  Baseline (n = 14) | 4.0 (1.0)
  Change at Month 12 (n = 14) | 4.0 (1.0)
  Change at Month 24 (n = 14) | 2.5 (1.3)
  Change at Month 36 (n = 12) | 1.8 (1.1)

5. Secondary Outcome: Height
Description: Height was measured using a wall mounted device (example, Harpenden stadiometer). The standing height of the participant was measured two times and the mean of these measurements was recorded.
Time Frame: Baseline, Month 12, Month 24, Month 36
Population: ITT set included all participants who received at least 1 dose of study medication and had at least 1 evaluation of height after start of study medication. Here "n" signifies those participants evaluated at that time point.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Genotonorm
Number analyzed (Participants) | 44
cm
  Baseline (n = 44) | 123.9 (17.3)
  Month 12 (n = 39) | 130.3 (17.5)
  Month 24 (n = 39) | 137.8 (16.9)
  Month 36 (n = 27) | 143.5 (15.8)

6. Secondary Outcome: Change From Baseline in Height at Month 12, Month 24 and Month 36
Description: as for outcome 5
Time Frame: Baseline, Month 12, Month 24, Month 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Genotonorm
Number analyzed (Participants) | 39
cm
  Change at Month 12 (n = 39) | 7.7 (2.1)
  Change at Month 24 (n = 39) | 14.9 (3.4)
  Change at Month 36 (n = 27) | 22.3 (3.7)

7. Secondary Outcome: Mean Height Standard Deviation Score (SDS) for Chronological Age (CA)
Description: Height was measured using a wall mounted device (example, Harpenden stadiometer). The standing height of the participant was measured two times and the mean of these measurements was recorded. Height SDS CA Yx = (height Yx - reference mean for CA Yx) / reference SD for CA Yx. Height in SDS was calculated using Sempe reference means and SD for height. CA calculated as integer (Date of height measurement-Date of birth)/365.25*12. SDS indicates how similar the participant was to the reference population.
Time Frame: Baseline, Month 12, Month 24, Month 36
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Genotonorm
Number analyzed (Participants) | 44
SDS
  Baseline (n = 44) | -2.84 (0.91)
  Month 12 (n = 39) | -2.42 (0.98)
  Month 24 (n = 39) | -2.09 (1.08)
  Month 36 (n = 27) | -1.72 (0.96)

8. Secondary Outcome: Change From Baseline in Height Standard Deviation Score (SDS) for Chronological Age (CA) at Month 12, Month 24 and Month 36
Description: Change in height SDS CA was derived by subtracting height SDS CA at baseline from Yx value. Height SDS CA (for both baseline and Yx) = (height - reference mean for CA)/reference SD for CA. Height in SDS was calculated using Sempe reference means and SD for height. CA calculated as integer (Date of height measurement - Date of birth)/365.25*12. SDS indicates how similar the participant was to the reference population.
Time Frame: Baseline, Month 12, Month 24, Month 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Genotonorm
Number analyzed (Participants) | 39
SDS
  Change at Month 12 (n = 39) | 0.41 (0.42)
  Change at Month 24 (n = 39) | 0.81 (0.60)
  Change at Month 36 (n = 27) | 1.03 (0.62)

9. Secondary Outcome: Mean Height Standard Deviation Score (SDS) for Bone Age (BA)
Description: Height SDS BA Yx = (height Yx - reference mean for BA Yx) / reference SD for BA Yx. Height in SDS was calculated using Sempe reference means and SD for height. BA was estimated locally using an X-ray from the left wrist and hand. SDS indicates how similar the participant was to the reference population.
Time Frame: Baseline, Month 12, Month 24, Month 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Genotonorm
Number analyzed (Participants) | 35
SDS
  Baseline (n = 35) | -0.71 (1.52)
  Month 12 (n = 32) | -0.55 (1.68)
  Month 24 (n = 32) | -0.49 (1.77)
  Month 36 (n = 20) | -0.30 (1.46)

10. Secondary Outcome: Change From Baseline in Height Standard Deviation Score (SDS) for Bone Age (BA) at Month 12, Month 24 and Month 36
Description: Change in height SDS BA was derived by subtracting height SDS BA at baseline from Yx value. Height SDS BA (for both baseline and Yx) = (height-reference mean for BA)/reference SD for BA. Height in SDS was calculated using Sempe reference means and SD for height. BA was estimated locally using an X-ray from the left wrist and hand. SDS indicates how similar the participant was to the reference population.
Time Frame: Baseline, Month 12, Month 24, Month 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Genotonorm
Number analyzed (Participants) | 28
SDS
  Change at Month 12 (n = 28) | -0.05 (1.04)
  Change at Month 24 (n = 27) | 0.06 (1.36)
  Change at Month 36 (n = 17) | 0.05 (1.32)

11. Secondary Outcome: Change From Baseline in Annual Growth Rate Standard Deviation Score (SDS) for Chronological Age (CA) at Month 12 and Month 24 in ITT Population
Description: Change in AGR SDS for CA derived by subtracting AGR SDS CA at baseline from Yx value. AGR at Yx= (height Yx-height Y[x-1])/([date of Yx-date of Y{x-1}]/365.25). AGR as SDS calculated using Sempe reference means and standard deviations (SD) for growth rate. AGR SDS CA (for both baseline and Yx)= (AGR-reference mean for growth rate CA)/reference SD for growth rate CA. CA calculated as integer (Date of height measurement-Date of birth)/365.25*12. SDS indicates how similar participant was to reference population.
Time Frame: Baseline, Month 12, Month 24
Population: ITT set included all participants who received at least 1 dose of study medication and had at least 1 evaluation of height after start of study medication. Here 'N' (Number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Genotonorm
Number analyzed (Participants) | 36
SDS
  Change at Month 12 (n = 36) | 3.23 (2.66)
  Change at Month 24 (n = 35) | 2.62 (2.05)

12. Secondary Outcome: Change From Baseline in Annual Growth Rate Standard Deviation Score (SDS) for Chronological Age (CA) at Month 12 and Month 24 in PP Population
Description: as for outcome 1
Time Frame: Baseline, Month 12, Month 24
Population: PP analysis set included all participants in the ITT set without a major protocol violation. Here 'N' (Number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Genotonorm
Number analyzed (Participants) | 14
SDS
  Change at Month 12 (n = 14) | 4.40 (2.12)
  Change at Month 24 (n = 14) | 2.97 (1.68)

13. Secondary Outcome: Mean Growth Rate Standard Deviation Score (SDS) for Bone Age (BA)
Description: AGR at Yx was derived by subtracting AGR at baseline from Yx value. AGR was calculated each year and rescaled to 1 year if the interval between Yx and Y[x-1] was not 365 days, as long as a participant remained in the study. AGR at Yx = [height Yx-height Y{x-1}] / ([date of Yx - date of Y{x-1}] /365.25). GR in SDS was calculated using Sempe reference means and SD for growth. BA was estimated locally using an X-ray from the left wrist and hand. SDS indicates how similar the participant was to the reference population.
Time Frame: Month 12, Month 24, Month 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Genotonorm
Number analyzed (Participants) | 28
SDS
  Month 12 (n = 28) | 1.06 (1.57)
  Month 24 (n = 25) | 0.46 (1.15)
  Month 36 (n = 19) | -0.01 (1.19)

14. Secondary Outcome: Body Mass Index (BMI)
Description: BMI was used to measure body fat based on height and weight. It was calculated as body weight (kilogram) divided by the height (meter) squared.
Time Frame: Baseline, Month 12, Month 24, Month 36
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)
Arm/Group | Genotonorm
Number analyzed (Participants) | 44
kilogram per square meter (kg/m^2)
  Baseline (n = 44) | 16.57 (2.37)
  Month 12 (n = 39) | 16.96 (2.64)
  Month 24 (n = 39) | 17.59 (2.69)
  Month 36 (n = 27) | 17.67 (2.08)

15. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) at Month 12, Month 24 and Month 36
Description: as for outcome 14
Time Frame: Baseline, Month 12, Month 24, Month 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Genotonorm
Number analyzed (Participants) | 39
kg/m^2
  Change at Month 12 (n = 39) | 0.52 (1.01)
  Change at Month 24 (n = 39) | 1.30 (1.35)
  Change at Month 36 (n = 27) | 1.89 (1.61)

16. Secondary Outcome: Change From Baseline in Bone Age (BA) at Month 12, Month 24 and Month 36
Description: BA was estimated locally using an X-ray from the left wrist and hand.
Time Frame: Baseline, Month 12, Month 24, Month 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Genotonorm
Number analyzed (Participants) | 40
years
  Baseline (n = 40) | 8.70 (3.28)
  Change at Month 12 (n = 28) | 1.69 (0.90)
  Change at Month 24 (n = 28) | 2.60 (0.97)
  Change at Month 36 (n = 21) | 4.04 (1.09)

17. Secondary Outcome: Ratio of Bone Age (BA) to Chronological Age (CA)
Description: BA was estimated locally using an X-ray from the left wrist and hand. CA at the date of corresponding X-ray (Date of X-ray - Date of birth)/365.25. Ratio of BA/CA at each annual study visit was calculated.
Time Frame: Baseline, Month 12, Month 24, Month 36
Population: ITT set included all participants who received at least 1 dose of study medication and had at least 1 evaluation of height after start of study medication. Here 'N' (Number of participants analyzed) signifies those participants who were evaluable for this measure and "n" signifies those participants evaluated at that time point.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Genotonorm
Number analyzed (Participants) | 40
ratio
  Baseline (n = 40) | 0.79 (0.15)
  Month 12 (n = 30) | 0.83 (0.15)
  Month 24 (n = 32) | 0.85 (0.12)
  Month 36 (n = 23) | 0.89 (0.14)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Genotonorm
Serious Adverse Events (participants affected / at risk) | 4/46
Other Adverse Events (participants affected / at risk) | 21/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Genotonorm (N=46)
Cryptorchism (Congenital, familial and genetic disorders) | 1
Laryngitis (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Weight decreased (Investigations) | 1
Histiocytosis haematophagic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Genotonorm (N=46)
Diarrhoea (Gastrointestinal disorders) | 2
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 2
Tracheitis (Infections and infestations) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Ammonia increased (Investigations) | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1
Insulin resistance (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Knee deformity (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Rickets (Musculoskeletal and connective tissue disorders) | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 5
Loss of consciousness (Nervous system disorders) | 1
Abnormal behaviour (Psychiatric disorders) | 1
Encopresis (Psychiatric disorders) | 1
Enuresis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1
Ear tube insertion (Surgical and medical procedures) | 1
Haematoma (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.